CLINICAL TRIAL: NCT07286097
Title: The Effect of Artistic Activities on Anxiety, Spiritual Well-Being, Hope, and Vital Signs in Patients Undergoing Abdominal Surgery: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Eda Ayten Kankaya, Asst. Prof., Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 9711-GOA
Record Dates: First submitted 2025-11-20; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-07

CONDITIONS: This Study Evaluates the Effect of Artistic Activities on Anxiety, Spiritual Well-being, Hope, and Vital Signs in Abdominal Surgery Patients
Keywords: Abdominal Surgery; Spiritual Well-being; Art Therapy
MeSH Terms: interventions — Breathing Exercises

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Art group (Experimental): mandala group
  Interventions: Behavioral: Art activities
- Control group (Active Comparator): deep breathing exercises
  Interventions: Behavioral: breathing exercises

INTERVENTIONS:
Behavioral: Art activities — In the study, pre-tests and post-tests were administered to patients in the experimental and control groups by the first researcher in the patients' rooms. The pre-test data for the study will be collected using the "Patient Diagnosis Form," "Vital Signs Form," "Visual Analog Anxiety Scale," "Spiritual Well-Being Scale," and "State Hope Scale" through face-to-face interviews lasting an average of 10 minutes. After the data is collected, the experimental group will participate in art activities from the body and mind therapy group, while the control group will perform breathing exercises. Final test data will be collected 10 minutes after the activities are completed.
  Arms: Art group
Behavioral: breathing exercises — the control group will perform breathing exercises
  Arms: Control group

SUMMARY:
The surgical process can cause high levels of anxiety and stress in patients, and abdominal surgery is particularly anxiety-provoking due to the risk of severe pain and complications. Artistic activities can be an effective complementary method for reducing anxiety and improving mental well-being and hope levels in individuals. Studies have shown that activities such as music therapy and visual arts have positive effects on pain, anxiety, and vital signs in surgical patients. This randomized controlled trial aims to evaluate the effects of artistic activities on anxiety, spiritual well-being, hope, and vital signs in patients undergoing abdominal surgery. The research will be conducted on patients undergoing abdominal surgery at the Department of General Surgery at Dokuz Eylül University. The data collection tools used will be the "Patient Assessment Form," "Vital Signs Form," "Visual Analog Anxiety Scale," "Spiritual Well-Being Scale," and "State Hope Scale." The intervention group will participate in mandala coloring as an artistic activity, while the control group will perform breathing exercises. Data analysis will be conducted using the SPSS 29.0 software package. Descriptive and analytical statistics will be used in the data analysis. The results of the study will determine the effect of artistic activities performed on abdominal surgery patients in the preoperative period on anxiety, spiritual well-being, hope, and vital signs. Based on the effectiveness of preoperative artistic activities in clinical use, a decision will be made as to whether they are useful in preparing patients for surgery in the preoperative period.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years of age or older

  * Be scheduled to undergo elective abdominal surgery (stomach, esophagus, colorectal, hepatobiliary)
  * Be conscious and able to communicate
  * Be willing to participate in the study

Exclusion Criteria:

* Patients requiring emergency abdominal surgery

  * Patients with chronic psychiatric disorders
  * Patients with severe cognitive impairment
  * Patients with severe hearing or vision loss
  * Patients requiring intensive care
  * Patients with degenerative brain disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2025-05-07 (Actual); Primary Completion 2025-08-07 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
anxiety | Baseline (pre-test), before the intervention - assessed once immediately prior to the intervention.
  Anxiety levels will be measured using the Visual Analog Anxiety Scale (VAAS). The scale ranges from 0 to 10, where 0 indicates no anxiety and 10 indicates the highest possible anxiety. Higher scores represent worse anxiety. The baseline (pre-test) measurement will be obtained during a face-to-face interview prior to the intervention.
Spiritual Well-Being | Baseline (pre-test), before the intervention - assessed once immediately prior to the intervention.
  Spiritual well-being will be assessed using the Spiritual Well-Being Scale.It was developed by Daaleman and Frey (2004), and its Turkish validity and reliability study was conducted by Serbest and Şahin (2022). The scale consists of 12 items and two subscales (self-efficacy and life plan). Participants' responses are rated on a 5-point Likert-type response scale ranging from 1 = "Strongly agree" to 5 = "Strongly disagree." The total score of the scale ranges from 12 to 60. The baseline (pre-test) measurement will be obtained during a face-to-face interview prior to the intervention.
State Hope | Baseline (pre-test), before the intervention - assessed once immediately prior to the intervention.
  Hope levels will be assessed using the State Hope Scale. The scale consists of six items. Responses were collected using an 8-point Likert scale (1= Strongly disagree, 4= Somewhat disagree, 8= Strongly agree).

SECONDARY OUTCOMES:
Vital signs | Baseline (pre-test), before the intervention-assessed once immediately prior to the intervention.
  Vital signs will be assessed using the Patient Vital Signs Form, which includes blood pressure, pulse, respiratory rate, temperature, and pain level. Measurements will be obtained following standard clinical procedures during the baseline (pre-test) assessment prior to the intervention. Values will be interpreted according to established physiological reference ranges, and higher pain scores represent worse symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: NAzife Gamze Özer Özlü, Phd, Principal Investigator — Dokuz Eylul university Nursing Faculty
Locations (1):
- Dokuz Eylul University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol